CLINICAL TRIAL: NCT00935363
Title: Interplay Between Organic Anion Transporting Polypeptide (OATP) Transporters Transporters and CYP2C9 in Glyburide Pharmacokinetics (PK)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GlyburideOATP2C9
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: glyburide; pharmacokinetics; pharmacodynamics; drug interaction; Healthy Volunteers
MeSH Terms: interventions — Glyburide; Fluconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- glyburide + fluconazole (Experimental)
  Interventions: Drug: glyburide + fluconazole
- glyburide + rifampin (Experimental)
  Interventions: Drug: glyburide + rifampin
- glyburide (Active Comparator)
  Interventions: Drug: glyburide
- glyburide + fluconazole + rifampin (Experimental)
  Interventions: Drug: glyburide + fluconazole + rifampin

INTERVENTIONS:
Drug: glyburide — single oral dose
  Arms: glyburide
Drug: glyburide + fluconazole — single dose oral glyburide single dose iv fluconazole
  Arms: glyburide + fluconazole
Drug: glyburide + rifampin — single dose oral glyburide single dose iv rifampin
  Arms: glyburide + rifampin
Drug: glyburide + fluconazole + rifampin — single dose oral glyburide single dose iv fluconazole single dose iv rifampin
  Arms: glyburide + fluconazole + rifampin

SUMMARY:
The purpose of this study is to investigate if the drugs rifampin and fluconazole when given together increase the concentrations in the body of the oral diabetes medication glyburide.

DETAILED DESCRIPTION:
The purpose of this study is to find out if a drug interaction occurs when glyburide is taken with rifampin and fluconazole. Glyburide is an oral drug commonly used to lower blood glucose levels in diabetic patients. Rifampin is an antibiotic used to treat tuberculosis and a variety of other infections caused by certain germs called bacteria. Both drugs affect a protein found in your liver cells called organic anion transporting polypeptides (OATPs). This protein regulates drugs getting into and out of your body. Fluconazole is commonly used to treat fungal infections like candidiasis, urinary tract infections and a variety of other infections caused by fungi. It interacts with glyburide by affecting your body's ability to breakdown glyburide. Since both rifampin and fluconazole play a role in the way glyburide enters and remains active in the body, we want to find out what effect taking the three drugs together has on the level of glyburide in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam and laboratory evaluations;
* BMI between 18.5 - 30 kg/m2;
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or OTC medications (except acetaminophen);
* Subjects must be able to maintain adequate birth control during the study independent of hormonal contraceptive use;
* Be able to provide written informed consent and comply with requirements of the study;
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until completion of the entire study;
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 6pm the night before a study day until completion of that study day;
* Fast from food and beverages at least 8 hours prior to medication dosing;
* Be able to read, speak and understand English

Exclusion Criteria:

* Subjects on prescription or chronic over-the counter medications (including hormonal contraceptives);
* Subjects with known allergy to glyburide and/or rifampin and/or fluconazole;
* Subjects who are not homozygous for CYP2C9 *1 (known poor metabolizers);
* Subjects with liver failure or LFTs >2x upper limit of normal;
* Subjects with clinically significant elevations in SCr, BUN or other screening laboratory tests as determined by study physician;
* Subjects with Hct <30 mg/dL;
* Subjects who smoke tobacco;
* Subjects with ongoing alcohol or illegal drug use;
* Subjects who are pregnant, lactating or attempting to conceive;
* Subjects unable to maintain adequate birth control during the study;
* Subjects unable to follow protocol instructions or protocol criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Drug Plasma Levels | 24 hours

SECONDARY OUTCOMES:
Blood sugar levels | 24 hours